CLINICAL TRIAL: NCT02962401
Title: An Open Label Non-randomized Phase II Study Exploring "Chemo-free " Treatment Association With Idelalisib + Obinutuzumab in Patient With Relapsed/Refractory Waldenstrom's Macroglobulinemia
Brief Title: Efficacity of Idelalisib and Obinutuzumab in Patient With Relapsed Refractory Waldenstrom's Macroglobulinemia
Acronym: RemodelWM3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RemodelWM3
Record Dates: First submitted 2016-10-26; First posted 2016-11-11 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — obinutuzumab; idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Idelalisib and Obinutuzumab (Experimental): 6 cycles of Idelalisib and Obinutuzumab
  Cycle 1 :
  Idelalisib 150 mg x 2 p.o. day 1 to 28 Obinutuzumab 1000mg I.V. (2 parts) 100mg day 1 and 900mg day 2 day 1, 8 and 15
  Cycle 2 - 6 :
  Idelalisib 150 mg x 2 p.o. day 1 to 28 Obinutuzumab 1000mg I.V. day 1
  Consolidation Idelalisib alone 150 mg twice a day until day 672 = 2 years after the beginning of the treatment
  Interventions: Drug: Obinutuzumab; Drug: Idelalisib

INTERVENTIONS:
Drug: Obinutuzumab — 6 cycles every 28 days Cycle 1 :Obinutuzumab 1000mg I.V.(2 parts) 100mg day 1 and 900mg day 2 day 1, 8 and 15
  Cycle 2 - 6 :
  Obinutuzumab 1000mg I.V.day 1
  Other Names: GA101
Drug: Idelalisib — 6 cycles every 28 days
  Cycle 1 :
  Idelalisib 150 mg x 2 p.o. day 1 to 28 Cycle 2 - 6 Idelalisib 150 mg x 2 p.o. day 1 to 28 Consolidation Idelalisib alone 150 mg twice a day until day 672 = 2 years after the beginning of the treatment
  Other Names: Zydelig

SUMMARY:
Prospective national multicenter open label phase II Remodel WM3 trial

DETAILED DESCRIPTION:
An Open Label non-randomized Phase II Study exploring chemo-free treatment association with Idelalisib and Obinutuzumab in Patient with relapsed refractory Waldenstrom's Macroglobulinemia

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Confirmed CD20 positive WM, according to the recommendations of the 2nd Workshop on WM.
* Presence of at least one criterion for initiation of therapy, according to the 2nd Workshop on WM.
* Recurrent fever, night sweats, weight loss, fatigue
* Hyperviscosity
* Lympadenopathy which is either symptomatic or bulky more or equal to 5cm in maximum diameter
* Symptomatic hepatomegaly and/or splenomegaly
* Symptomatic organomegaly and/or organ or tissue infiltration
* Peripheral neuropathy due to WM
* Symptomatic cryoglobulinemia
* Cold agglutinin anemia
* Immune hemolytic anemia and/or thrombocytopenia
* Nephropathy related to WM
* Amyloidosis related to WM
* Hemoglobin less or equal than 10g dL
* Platelet count less than 100 109 L
* Prior treatment for WM comprising at least one regimen containing a therapeutic anti CD20 monoclonal antibody rituximab administered for more or equal than 2 doses of antibody treatment and or a therapeutic chemotherapy, alkylating agent, purine analogue, bendamustine administered for more or equal than 2 cycles of treatment
* Patients may be either relapsing progressing at least 6 months after the last administration of first line or subsequent treatment or refractory progressing on or within 6 months of first line or subsequent treatment
* Number of prior regimens per lines 1 to 3
* Life expectancy more than 3 months.
* ECOG less or equal than 2.
* Meet the following pretreatment laboratory criteria at the screening visit conducted within 28 days of study enrollment:

  * ASAT 2.5 times the upper limit of institutional laboratory normal value.
  * ALAT 2.5 times the upper limit of institutional laboratory normal value.
  * Total bilirubin 1.5 times the upper limit of institutional laboratory normal value unless clearly related to the disease or Gilbert syndrome
  * Calculated or measured creatinin clearance by MDRD 40 mL minute.
* Premenopausal fertile females must agree to use a highly effective method of birth control for the duration of the therapy up to 6 months after end of therapy.
* A highly effective method of birth control is defined as those which result in a low failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.
* Men must agree not to father a child for the duration of therapy and 6 months after and must agree to advice a female partner to use a highly effective method of birth control.
* Voluntary written informed consent before carrying out any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Prior treatment with phosphatidylinositol 3 kinase PI3K inhibitors including idelalisib or GA101
* History of anaphylactic reaction following exposure to humanized monoclonal antibodies
* Previous allogeneic transplantation
* Treatment with any other investigational agent or participating in another trial within 30 days prior to entering this study
* History of other malignancy or chemotherapy radiotherapy for any neoplastic disease other than WM prior to the study.

  * EXCEPTION: History of malignancy except basal cell carcinoma of the skin, in situ carcinoma of breast or cervix treated surgically with curative intent, or any malignancy that has been in CR for 5 years at minimum, or as deemed appropriate for inclusion in the trial as per approval by the investigator
* Medical condition requiring the long-term estimated to be more than one month use of oral corticosteroids.
* Patients with signs of bacterial, viral or fungal infection
* Preexisting hepatic enzyme elevation ASAT, ALAT
* CMV PCR or antigenemia testing positive
* Known history of drug induced liver injury, chronic active hepatitis C HCV, chronic active hepatitis B HBV, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, on-going extra-hepatic obstruction caused by cholelithiasis, cirrhosis of the liver or portal hypertension
* HIV antibody positive
* Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb): Patients with presence of HBcAb, but absence of HBsAg, are eligible if hepatitis B virus (HBV) DNA is undetectable (< 20 IU). Patients with positive serology should be referred to a hepatologist or gastroenterologist before start of treatment and should be monitored and managed following local standards to prevent hepatitis reactivation. Furthermore transaminases and HBV DNA quantification must be tested at weeks 4 and 8 after treatment start. Then transaminases must be tested at week 12 of treatment start.
* Preexisting pulmonary disease
* Known history of drug induced pneumonitis
* On-going inflammatory bowel disease
* Women who are pregnant. Women who are breast-feeding and do not consent to discontinue breast-feeding Women of childbearing age who are not willing to use effective anti-conceptive methods for the duration of the study and 6 months after end of therapy
* Concurrent severe diseases which exclude the administration of therapy:
* Heart insufficiency NYHA grade III IV, LVEF < 50% and or RF <30%, myocardial infarction within the past 6 months prior to study
* Severe chronic obstructive lung disease with hypoxemia
* Severe diabetes mellitus
* Hypertension difficult to control
* Cerebral dysfunction
* Richter's syndrome
* Cardiac amyloidosis
* Any of the following laboratory abnormalities, if not related to lymphoma:
* Absolute neutrophils count <1.5 x 109/L if not result of a bone marrow infiltration Platelet count <75 x 109/L if not result of a bone marrow infiltration.
* Central Nervous System involvement by lymphoma
* Vaccination with live vaccines within 28 days prior to study entry
* Hypersensitivity to the active substance or to any of the excipients listed on part 6.1 of GAZYVARO and ZYDELIG SmCP
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* No consent for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician about study participation
* Patient with mental deficiency preventing proper understanding of the requirements of treatment
* Person major under law control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 8 years
  From date of registration until the date of first documented progression or date of death

SECONDARY OUTCOMES:
Overall response rates (ORR) | Month 8
  treatment response
Duration of response (RD) | 7 years and 4 months
  from end of induction to the date of progression, relapse or death
Time to treatment failure (TTF) | through study completion, an average of 8 years
  time from start of induction to stable disease, progression or death from any cause
Time to next treatment (TTNT) | through study completion, an average of 8 years
  time from start of induction day 1 cycle 1 to time of the next treatment for progression or relapse

CONTACTS AND LOCATIONS:
Overall Officials: Adeline LHERMITTE, Mrs, Study Director — French Innovative Leukemia Organisation
Locations (1):
- Project manager, Tours, France

IPD SHARING:
Plan to Share IPD: Yes
E CRF

REFERENCES:
- [Derived] Tomowiak C, Poulain S, Nudel M, Feugier P, Herbaux C, Mahe B, Morel P, Aurran T, Tournilhac O, Lepretre S, Assaad S, Villemagne B, Casasnovas O, Lhermitte A, Roos-Weil D, Torregrosa-Diaz J, Chevret S, Leblond V; on the behalf of the FILO group. Six-year follow-up of phase II study exploring chemo-free treatment association with idelalisib and obinutuzumab in symptomatic relapsed/ refractory patients with Waldenstrom's macroglobulinemia. Ann Hematol. 2025 Jan;104(1):685-690. doi: 10.1007/s00277-024-06076-1. Epub 2024 Nov 5. PMID 39499299
- [Derived] Tomowiak C, Poulain S, Herbaux C, Perrot A, Mahe B, Morel P, Aurran T, Tournilhac O, Lepretre S, Assaad S, Villemagne B, Casasnovas O, Nollet D, Roos-Weil D, Chevret S, Leblond V. Obinutuzumab and idelalisib in symptomatic patients with relapsed/refractory Waldenstrom macroglobulinemia. Blood Adv. 2021 May 11;5(9):2438-2446. doi: 10.1182/bloodadvances.2020003895. PMID 33961019
- See also: FILO internet site — http://www.filo-leucemie.org